CLINICAL TRIAL: NCT06026228
Title: Effects of Oral Intake of the Probiotic Limosilactobacillus Reuteri on Plasma Chlordecone (Kepone) Concentrations (Chlordeconemia) in Individuals Environmentally Exposed to the Organochlorine Pesticide in Martinique : an Exploratory Pilot Study
Brief Title: Effects of Probiotic Oral Intake on Plasma Chlordecone (Kepone) Concentrations in Individuals Environmentally Exposed to Pesticide in Martinique.
Acronym: CHLOR-DETOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: BioGaia AB (Industry); University Hospital, Limoges (Other); Regional Health Agency, Martinique (Unknown); Biological Resource Centre, Martinique (Unknown); Reims University hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21_RIPH3-08; 2021-A02293-38 (Other: French National Medicines and Health Products safety Agency)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Chlordecone (Kepone) Toxicity
Keywords: Chlordecone toxicity; Probiotics; Gut elimination; entero-hepatic cycle; plasma level concentration

STUDY DESIGN:
Intervention Model Description: This is a study in two parallel groups of equal numbers: control group (placebo) and experimental group (probiotic).
  The control group will receive daily a placebo capsule per os at mealtime (just before or after) for a period of 6 months.
  The experimental group will receive daily per os one capsule of BioGaia® Gastrus probiotic , taken at mealtime (just before or after) for a period of 6 months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking will be carried out by the hospital pharmacy, which will dispense the appropriate batches to the team, following the randomisation list established by the Methodology and Data Management Centre.
  The hospital pharmacy, will keep a batch matching table, which will be made available to the vigilance unit and the Methodology and Data Management Centre.
  Masking will be maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The control group will receive daily a placebo capsule per os at mealtime (just before or after) for a period of 6 months
  Interventions: Other: Placebo
- Experimental group (Experimental): The experimental group will receive daily per os one capsule of BioGaia® Gastrus probiotic (combination of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475) dosed at 108 colony forming units (CFU)/day (distributed by the laboratory PEDIACT France), taken at mealtime (just before or after) for a period of 6 months
  Interventions: Dietary Supplement: Limosilactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri — The BioGaia® Gastrus probiotic capsule contains the following components: L. reuteri DSM 17938, L. reuteri ATCC PTA 6475) at 10^8 CFU*/day, fully hydrogenated palm oil; ascorbic acid; tangerine flavour and mint flavour.
  *Colony forming Unit
  Other Names: BioGaïa® Gastrus
  Arms: Experimental group
Other: Placebo — The placebo capsules have the same external appearance and composition as the BioGaia® Gastrus Limosilactobacillus reuteri probiotic capsule (combination of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475), but without the active ingredient.
  Arms: Control group

SUMMARY:
The CHLOR-DETOX study is a single-centre, double-blind, prospective, interventional, controlled, exploratory pilot study on subjects environmentally exposed to the organochlorine pesticide (kepone or chlordecone, CLD) in the French Caribbean (Martinique island). To our best knowledge, it is the first clinical trial in such subjects evaluating the potential effect of oral probiotic intake (Limosilactobacillus reuteri) on the reduction of CLD plasma levels (chlordeconemia) and fecal excretion, thus concurring to the reduction of CLD toxicity in study subjects.

DETAILED DESCRIPTION:
The research question focuses on the ability of the probiotic Limosilactobacillus reuteri Gastrus (combination of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475 from the BioGaia® company) to reduce CLD toxicity in subjects exposed to this pesticide. In particular, the investigators are interested in whether the oral prescription of Limosilactobacillus reuteri reduces plasma levels of CLD by increasing the fecal excretion of the deconjugated form of CLD. This research hypothesis is based on the presence of a hydrolase activity (glucuronidase) in Limosilactobacillus reuteri that allows the deconjugation of glucuronide derivatives (De Boever et al 2000; Cardona et al. 2002; Martoni et al 2008). Limosilactobacillus reuteri is the probiotic with the highest hydrolase activity. The combination of Limosilactobacillus reuteri DSM 17938 and Limosilactobacillus reuteri ATCC PTA 6475 (BioGaia® Gastrus) is currently the best possible formulation for optimal hydrolase activity (unpublished data from BioGaia® laboratory). The investigators also hypothesize that the increase in CLD elimination by the digestive tract through the use of Limosilactobacillus reuteri avoids the appearance of side effects encountered during the prolonged use of classical bile salt sequestrants (e.g. QUESTAN).

The effects of oral prescription of Limosilactobacillus reuteri on plasma levels and faecal concentrations of CLD will be compared with a control group under placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older
* Seen in clinical toxicology consultation at the CHU of Martinique during the study period
* With an initial chlordeconemia > 1μg/L on a test less than 1 month old at the time of study inclusion
* Affiliated to a social security scheme
* Having received informed information on research
* Having freely given written and informed consent to participate in the research

Exclusion Criteria:

* History of cancer
* Recent infections less than 6 months old
* Known digestive diseases: chronic diarrhoea, ulcerative colitis, Crohn's disease, pancreatitis
* Digestive procedures less than 6 months old.
* Intrahepatic cholestasis less than 6 months old
* Extrahepatic cholestasis less than 6 months old
* Use of cholestyramine or ursodeoxycholic acid in the previous 3 months
* Consumption of food (non-ordinary yoghurt, etc.) or supplements (tablets, drops, capsules, etc.) containing L. reuteri or any other probiotic within the previous 2 weeks.
* Antibiotics taken in the previous 4 weeks.
* Immune deficiency secondary to a pathology (lymphoma, leukaemia) or medical treatment (immunosuppressant, corticoid, chemotherapy).
* Women who are unable to obtain contraception during the trial
* Persons referred to in articles L.1121-5, L.1121-7, L. 1121-8 of the Public Health Code:

  * Pregnant woman, parturient or breastfeeding mother
  * Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
  * Persons deprived of their liberty by a judicial or administrative decision,
  * Persons staying in a health or social care institution for purposes other than research
* Persons subject to psychiatric care under Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Chlordeconemia | 6 months
  Chlordeconemia measured by a gas chromatography/mass spectrometry (GC/MS) technique expressed in μg/L (analytical detection limit LDD of 0.05 μg/L - quantification limit LDQ of 0.1 μg/L)
  The relative change in chlordeconemia between T0 and T6 months will be compared between the group of patients treated with the BioGaia® Gastrus probiotic and the group of patients treated with placebo.
  This relative variation will be calculated as the ratio of the difference in chlordeconemia T0 -T6mois to the initial chlordeconemia at T0.

SECONDARY OUTCOMES:
Chlordeconemia | 3 months
  Chlordeconemia measured by a gas chromatography/mass spectrometry (GC/MS) technique expressed in μg/L (analytical detection limit LDD of 0.05 μg/L - quantification limit LDQ of 0.1 μg/L
  The relative change in chlordeconemia between T0 and T3months will be compared between the BioGaia® Gastrus probiotic treated group and the placebo treated group.
  This relative variation will be calculated as the ratio of the difference in chlordeconemia T0 -T3months to the initial chlordeconemia at T0.
Variation of chlordeconemia | 6 months
  The relative variation of chlordeconemia from T0 to T6 months in each group of patients (probiotic group, placebo group) will be described. The plasma half-life values of CLD, expressed in months, will be determined for each group.
concentration of CLD in the stool | 6 months
  The concentration of CLD in the stool at 3 months (T3 months) and 6 months (T6 months) will be measured using the same method described in the primary outcome (GC/MS technique). The relative changes in stool CLD concentration between T0 and T3mois and T0 and T6mois will be compared between the BioGaia® Gastrus probiotic treated group and the placebo treated group.
Variation of chlordecone concentration in stool | 6 months
  - The relative change in stool CLD concentration from T0 to T6months within each patient group (probiotic group, placebo group) will be described
Plasma total cholesterol concentrations | 6 months
  Plasma total cholesterol concentrations, measured by the reference technique (ultracentrifugation followed by heparin-manganese precipitation and then quantification by the Abell-Kendall method) at T0 , T3 months and T6 months will be described. The relative variations of plasma total cholesterol concentrations between T0 and T3months and T0 and T6months will be compared between the group of patients treated with the BioGaia® Gastrus probiotic and the group of patients treated with placebo.
Clinical tolerance to BioGaia® Gastrus probiotic or placebo | 6 months
  Treatments will be assessed by adverse event reporting and based on a standardised and internationally recognised toxicity table for adults.
  This tolerance will be assessed by a telephone interview at T1 month, T2 months, T4 months and T5 months, as well as during face-to-face follow-up visits at T3months and T6months .

CONTACTS AND LOCATIONS:
Overall Officials: DABOR RESIERE, Professor, Principal Investigator — University Hospital of Martinique
Locations (1):
- Centre Hospitalier Universitaire de Martinique - Hôpital Pierre ZOBDA QUITMAN, Fort-de-France, France, Martinique

IPD SHARING:
Plan to Share IPD: No